CLINICAL TRIAL: NCT01908660
Title: Hepatic Safety of Currently Used Antiretroviral Regimens in HIV-infected Patients With Chronic Hepatitis B and/or Hepatitis C Under Real Life Conditions: The HEPAVIR HEPATIC SAFETY Cohort.
Brief Title: Hepatic Safety of Currently Used Antiretroviral Regimens in Patients With Chronic Hepatitis Under Real Life Conditions
Status: Completed | Type: Observational
Sponsor: Valme University Hospital (Other)
Collaborators: Hospital Universitario Virgen de la Victoria (Other); Hospital Universitario Reina Sofia de Cordoba (Other Government); Hospital Torrecárdenas (Unknown); Hospital de la Línea de la Concepción (Unknown); Hospital Poniente (Unknown); Hospital Universitario Virgen Macarena (Other); Complejo Hospitalario de Especialidades Juan Ramón Jimenez (Other)
Responsible Party: Principal Investigator, Karin Neukam, PhD, Valme University Hospital
Other Study IDs: SEG-HEP-2007
Record Dates: First submitted 2013-06-28; First posted 2013-07-26 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Human Immunodeficiency Virus; Hepatitis B, Chronic; Hepatitis C, Chronic
Keywords: HIV; hepatitis C virus; hepatitis B virus; antiretroviral drugs; nucleos(t)ide reverse transcriptase inhibitors; non-nucleos(t)ide reverse transcriptase inhibitors; protease inhibitors; integrase inhibitors; entry inhibitors; transaminase elevations; alanine aminotransferase; aspartate aminotransferase; bilirubin elevations; hepatic fibrosis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hepatitis B, Chronic; Hepatitis C, Chronic; Hepatitis C; Hepatitis B; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Antiretroviral drugs: Pre-treated or treatment-naive HIV-infected patients with chronic hepatitis B and/or chronic hepatitis C who change an existing antiretroviral regimen or who start a new regimen.
  Interventions: Drug: antiretroviral drugs

INTERVENTIONS:
Drug: antiretroviral drugs — zidovudine lamivudine emtricitabine abacavir tenofovir nevirapine efavirenz etravirine rilpivirine lopinavir atazanavir fosamprenavir darunavir raltegravir maraviroc ritonavir

SUMMARY:
The purpose of this study is to compare the liver toxicity in HIV-infected patients with chronic hepatitis B and/or hepatitis C, who start a new antiretroviral drug regimen, as well as the influence of the degree of pre-existing liver fibrosis on the incidence of liver toxicity.

DETAILED DESCRIPTION:
In the last years, various clinical trials and studies have evaluated the incidence of hepatic toxicity (HT) associated with the commonly used antiretroviral drugs in the HIV/hepatitis C virus (HCV)-infected population. Unfortunately, clinical trials that compared hepatic safety of these antiretrovirals include a low number of coinfected patients (van Leth 2004, Molina 2010, Ortiz 2008, Rockstroh 2012). According to recent cohort studies, rates of grade 3 or 4 transaminase elevations (TE) observed in patients receiving ritonavir-boosted protease inhibitors PI/r as lopinavir (LPV/r), atazanavir (ATV/r), fosamprenavir (FPV/r) and darunavir (DRV/r) are similar to those observed in individuals that receive efavirenz (EFV) or raltegravir (RAL) (Pineda 2008, Palacios 2006, Macías 2011, Neukam 2011). However, this conclusion may not be exact due to methodological problems. In this context, currently available data on severe TE are derived from cohort studies that were conducted in different populations, with distinct methods and/or data that was collected retrospectively.

Little information is available on whether the stage of liver damage influences the incidence of HT caused by antiretroviral drugs. Although two studies found an association between advanced fibrosis and higher rates of TE (Aranzabal 2005, Mira 2006), data obtained by further studies are contradictory (Pineda 2008, Palacios 2006, Macías 2011, Neukam 2011) and there are still open questions. Thus, the number of cirrhotic patients is considerably small in these cohorts, however, cirrhosis represents an important comorbidity in HIV. In these individuals, plasmatic concentrations of antiretroviral drugs could reach toxic levels which would be reflected in TE (Barreiro 2007).

Therefore, studies conducted in the same population and with the same methodology are required in order to obtain precise and reliable information on hepatic safety of all commonly used antiretroviral drugs in the clinical practice. These findings could contribute to a better understanding of differences between antiretrovirals and could therefore improve the individualization of antiretroviral therapy in individuals with chronic hepatitis B and/or C. Therefore, the HEPAVIR group of the Andalusian Society of Infectious Diseases (SAEI) has established a prospective cohort: The HEPAVIR Cohort.

Hypothesis: The incidence of severe TE associated with antiretroviral therapy in the clinical practice in hepatitis B virus and/or hepatitis C virus-coinfected patients could be different according to the administered drug.

Primary objective: To determine the incidence of grade 3 or 4 TE associated with antiretroviral therapy in the clinical practice in patients with viral hepatitis.

Secondary objectives:

* Identification of factors associated with grade 3 or 4 TE
* Analysis of the association between TE and pre-existing hepatic damage
* Evaluate the incidence of serious symptoms, including hepatic decompensations, acute fulminant hepatitis and death due to liver failure, associated with the antiretroviral drug
* Determination of the incidence of grade 3 or 4 bilirubin elevations associated with the antiretroviral drugs
* Evaluation of efficacy of the antiretroviral drugs used in the study

Scheduled visits: 0, 4, 12, 24, 36 and 48 weeks.

Definition of grade 3 or 4 laboratory abnormalities/data dictionary: Grade 3 transaminase elevations (TE) are considered when elevations between 5 and 10 times above the upper level of normality (ULN) are presented in patients with normal baseline levels of alanine-aminotransferase (ALT) and aspartate-aminotransferase (AST). Grade 4 TE are defined as ALT or AST values >10 times of the ULN. In patients with elevated baseline ALT or AST levels, 3.5- to 5-fold increase from baseline levels are considered grade 3 TE and >5-fold elevations grade 4 TE, respectively. Grade 4 total bilirubin elevations were defined as increases of total bilirubin ≥5 mg/dl.

Definition of hepatic fibrosis:

* advanced fibrosis: F3 as determined by liver biopsy or 11 kilopascals as determined by transient elastometry
* cirrhosis: F4 as determined by liver biopsy or 14.6 kilopascals as determined by transient elastometry

Variables collected within in the cohort:

* primary outcome variable: AST, ALT
* epidemiological variable: age, sex
* variables related to hepatitis C virus-infection: infection route, genotype, grade of hepatic fibrosis and method used for its determination, baseline Child-Pough-Index, previous hepatic decompensations
* variables related to HIV-infection: Centers for Disease Control and Prevention (CDC) category, HIV viral load, cluster of differentiation 4 (CD4) cell count, previous and new antiretroviral drugs
* analytical variables: platelets, cholesterol, bilirubin, gamma-glutamyltransferase (GGT), alkaline phosphatase
* clinical variables: alcohol intake
* time to TE
* percentage of patients who discontinued antiviral therapy due to TE

Quality assurance and data checks: Data will be obtained from controlled databases at the participating centers. Databases will be monitored and controlled by queries every six months. Descriptive statistics will be be applied in order to detect transcription errors.

Source data verification: not planned.

All grade 3 or 4 adverse events, as well as all unexpected events, will be reported to the Andalusian Center for Pharmacovigilance (Centro Andaluz de Farmacovigilancia, www.cafv.es).

A sample size of 500 is planned for this study.

Statistical analysis:

The outcome variables of this study will be the development of grade 3 or 4 transaminase elevations (TE) and grade 4 total bilirubin elevations (TBE) during follow-up. Comparative analyses of TE and TBE will be carried out between the different drug groups. Additionally, the relationship between the outcome variable and the following potential predictors will be assessed: age, sex, previous intravenous drug use, alcohol consumption, baseline ALT levels, baseline CD4 cell count, CDC category C, undetectable plasma HIV-RNA, HCV genotype, previous ART, type of drug, as well as significant fibrosis and cirrhosis at initiation of the new ART regimen. Continuous variables will be expressed as median [interquartile range (IQR)] and categorical variables as number [percentage; 95% confidence interval (CI)]. The density of incidence of grade 3-4 TE will be calculated as number of cases per 100 person-years of the follow-up. Continuous variables will be compared using the Student's t-test for normal distribution and the Mann-Whitney U-test otherwise, whereas the categorical variables will be analyzed applying the χ2-test or the Fisher's test, when applicable. The Wilcoxon Signed Rank test and the McNemar test will be applied to compare repeated measurements in continuous and categorical variables, respectively. Those factors that show an association in the univariate analysis with a p<0.2, as well as those with a biologically possible influence, will be entered into a logistic regression model in order to identify independent risk factors for grade 3-4 TE and grade 4 TBE. The adjusted odds ratio (AOR) and the respective 95% CI will be calculated. All p values <0.05 will be considered statistically significant. Data will be analysed using the SPSS statistical software package release 19.0 (SPSS Inc., Chicago, IL, USA) and STATA 9.0 (StataCorp LP, College Station, TX, USA).

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* HIV-1 infection as confirmed by ELISA and western blot
* Chronic HCV infection as confirmed by HCV antibodies in plasma, as well as a positive HCV viral load determined by polymerase chain reaction OR chronic hepatitis B infection as confirmed by HBsAg
* Treatment-naive or pretreated patients who start a new antiretroviral regimen that includes at least one drug that has not been received by the patient before
* At least one week of exposure to new regimen
* Liver biopsy or transient elastometry determination within 12 months prior to treatment initiation

Exclusion Criteria:

* Pregnancy
* Treatment against hepatitis C virus infection
* Presence of opportunistic infections, including tuberculosis, neoplasia, autoimmune diseases. Patients receiving primary or secondary chemotherapy against an opportunistic process are not included.
* Any liver disease of vascular, metabolic, biliary, autoimmune or tumoral origin
* Patients who are not able to provide written informed consent to participate in the study
* Lack of scheduled clinical visits including blood analysis throughout study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen at the infectious disease unit of a terciary care center
Sampling Method: Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2007-01; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Incidence of grade 3 or 4 transaminase elevations | one year

SECONDARY OUTCOMES:
Incidence of grade 3 or 4 bilirubin elevations | one year
Percentage of patients with undetectable HIV RNA at the end of follow-up | one year
CD4 cell count at the end of follow-up | one year

CONTACTS AND LOCATIONS:
Overall Officials: Karin I Neukam, PhD, Principal Investigator — Hospital Universitario de Valme
Locations (1):
- Hospital Universitario de Valme, Seville, Spain

REFERENCES:
- [Background] van Leth F, Phanuphak P, Ruxrungtham K, Baraldi E, Miller S, Gazzard B, Cahn P, Lalloo UG, van der Westhuizen IP, Malan DR, Johnson MA, Santos BR, Mulcahy F, Wood R, Levi GC, Reboredo G, Squires K, Cassetti I, Petit D, Raffi F, Katlama C, Murphy RL, Horban A, Dam JP, Hassink E, van Leeuwen R, Robinson P, Wit FW, Lange JM; 2NN Study team. Comparison of first-line antiretroviral therapy with regimens including nevirapine, efavirenz, or both drugs, plus stavudine and lamivudine: a randomised open-label trial, the 2NN Study. Lancet. 2004 Apr 17;363(9417):1253-63. doi: 10.1016/S0140-6736(04)15997-7. PMID 15094269
- [Background] Molina JM, Andrade-Villanueva J, Echevarria J, Chetchotisakd P, Corral J, David N, Moyle G, Mancini M, Percival L, Yang R, Wirtz V, Lataillade M, Absalon J, McGrath D; CASTLE Study Team. Once-daily atazanavir/ritonavir compared with twice-daily lopinavir/ritonavir, each in combination with tenofovir and emtricitabine, for management of antiretroviral-naive HIV-1-infected patients: 96-week efficacy and safety results of the CASTLE study. J Acquir Immune Defic Syndr. 2010 Mar;53(3):323-32. doi: 10.1097/QAI.0b013e3181c990bf. PMID 20032785
- [Background] Ortiz R, Dejesus E, Khanlou H, Voronin E, van Lunzen J, Andrade-Villanueva J, Fourie J, De Meyer S, De Pauw M, Lefebvre E, Vangeneugden T, Spinosa-Guzman S. Efficacy and safety of once-daily darunavir/ritonavir versus lopinavir/ritonavir in treatment-naive HIV-1-infected patients at week 48. AIDS. 2008 Jul 31;22(12):1389-97. doi: 10.1097/QAD.0b013e32830285fb. PMID 18614861
- [Background] Rockstroh J, Teppler H, Zhao J, Sklar P, Harvey C, Strohmaier K, Leavitt R, Nguyen BY. Safety and efficacy of raltegravir in patients with HIV-1 and hepatitis B and/or C virus coinfection. HIV Med. 2012 Feb;13(2):127-31. doi: 10.1111/j.1468-1293.2011.00933.x. Epub 2011 May 22. PMID 21599819
- [Background] Pineda JA, Santos J, Rivero A, Abdel-Kader L, Palacios R, Camacho A, Lozano F, Macias J; Liverey Study Investigator Team. Liver toxicity of antiretroviral combinations including atazanavir/ritonavir in patients co-infected with HIV and hepatitis viruses: impact of pre-existing liver fibrosis. J Antimicrob Chemother. 2008 Apr;61(4):925-32. doi: 10.1093/jac/dkn045. Epub 2008 Feb 14. PMID 18276600
- [Background] Palacios R, Vergara S, Rivero A, Aguilar I, Macias J, Camacho A, Lozano F, Garcia-Lazaro M, Pineda JA, Torre-Cisneros J, Marquez M, Santos J. Low incidence of severe liver events in HIV patients with and without hepatitis C or B coinfection receiving lopinavir/ritonavir. HIV Clin Trials. 2006 Nov-Dec;7(6):319-23. doi: 10.1310/hct0706-319. PMID 17197379
- [Background] Macias J, Neukam K, Portilla J, Iribarren JA, de Los Santos I, Rivero A, Marquez M, Delgado M, Tellez F, Merino D, Giner L, von Wichmann MA, Pineda JA; HEPRAL study team. Liver tolerance of raltegravir-containing antiretroviral therapy in HIV-infected patients with chronic hepatitis C. J Antimicrob Chemother. 2011 Jun;66(6):1346-50. doi: 10.1093/jac/dkr083. Epub 2011 Mar 10. PMID 21398295
- [Background] Aranzabal L, Casado JL, Moya J, Quereda C, Diz S, Moreno A, Moreno L, Antela A, Perez-Elias MJ, Dronda F, Marin A, Hernandez-Ranz F, Moreno A, Moreno S. Influence of liver fibrosis on highly active antiretroviral therapy-associated hepatotoxicity in patients with HIV and hepatitis C virus coinfection. Clin Infect Dis. 2005 Feb 15;40(4):588-93. doi: 10.1086/427216. Epub 2005 Jan 21. PMID 15712082
- [Background] Barreiro P, Rodriguez-Novoa S, Labarga P, Ruiz A, Jimenez-Nacher I, Martin-Carbonero L, Gonzalez-Lahoz J, Soriano V. Influence of liver fibrosis stage on plasma levels of antiretroviral drugs in HIV-infected patients with chronic hepatitis C. J Infect Dis. 2007 Apr 1;195(7):973-9. doi: 10.1086/512086. Epub 2007 Feb 20. PMID 17330787
- [Result] Neukam K, Mira JA, Ruiz-Morales J, Rivero A, Collado A, Torres-Cornejo A, Merino D, de Los Santos-Gil I, Macias J, Gonzalez-Serrano M, Camacho A, Parra-Garcia G, Pineda JA; SEGURIDAD HEPATICA Study Team of the Grupo HEPAVIR de la Sociedad Andaluza de Enfermedades Infecciosas (SAEI). Liver toxicity associated with antiretroviral therapy including efavirenz or ritonavir-boosted protease inhibitors in a cohort of HIV/hepatitis C virus co-infected patients. J Antimicrob Chemother. 2011 Nov;66(11):2605-14. doi: 10.1093/jac/dkr357. Epub 2011 Sep 7. PMID 21903660